CLINICAL TRIAL: NCT02611999
Title: The Effect of Paid Price Information on Image and Procedure Ordering Rates
Brief Title: Paid Price Information on Image and Procedure Ordering Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Atrius Health (Other)
Responsible Party: Principal Investigator, Alyna Chien, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P00011096
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Physicians' ordering behavior with price information

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Control (No Intervention): Physicians in this Arm received only a paper memo with a list of common imaging tests and procedures.
- Single Price (Experimental): Physicians in this Arm received a single median price in the electronic medical record at the time of ordering in addition to the paper memo.
  Interventions: Behavioral: Single median price information
- Paired Inside/Outside Prices (Experimental): Physicians in this Arm received two prices (the inside and outside price) in the electronic medical record at the time of ordering in addition to the paper memo.
  Interventions: Behavioral: Paired inside/outside price information

INTERVENTIONS:
Behavioral: Single median price information — Physicians in this Arm received a single median price in the electronic medical record at the time of ordering in addition to the paper memo.
  Arms: Single Price
Behavioral: Paired inside/outside price information — Physicians in this Arm received two prices (the inside and outside price) in the electronic medical record at the time of ordering in addition to the paper memo.
  Arms: Paired Inside/Outside Prices

SUMMARY:
The investigators' study seeks to explore the impact of price information on physicians' ordering behavior and care quality. The investigators will evaluate the impact of the physician price transparency initiative at Atrius Health (ATRIUS) on rate of overall procedure and test orders, clinically inappropriate orders, and appropriate orders. Ultimately, this study will help stakeholders understand the degree to which price information can help improve the value of healthcare.

DETAILED DESCRIPTION:
The investigators' study team worked with Atrius Health (ATRIUS) to design a physician price transparency (PPT) intervention aimed at providing primary and specialty care physicians with price information on commonly-ordered outpatient procedures (e.g., Pap smears, ECHOs, colonoscopies) and imaging tests (e.g., CTs and MRIs). The 2014 PPT intervention was built upon a pilot that ATRIUS conducted in 2010. Starting January 1, 2014, ATRIUS randomized its physicians to 3 different study arms, those receiving:

1. No price display for common outpatient procedures or imaging tests,
2. A single price for each procedure or test, or
3. A pair of prices for each procedure or test (that allowed physicians to compare prices that would be charged if the test was conducted at a facility within the ATRIUS network versus outside of it).

The mode for delivering this PPT intervention was ATRIUS' common electronic medical record (EMR), which all of its physicians use to place all orders related to outpatient procedures and imaging studies.

The investigators used a blocked randomized-controlled study design to quantitatively and qualitatively evaluate the effect of No, Single and Paired procedure and imaging test price information on: rate of overall procedure and test orders, clinically inappropriate orders, and appropriate orders.

The investigators used ATRIUS' administrative and EMR Data Repository to assess the quantitative outcomes proposed within this study. This repository contains the information the investigators need to block randomize at the practice level and to describe practices (e.g., size, location) and physicians (e.g., age, gender, specialty). It also captures all of the actions that physicians take when caring for patients (all orders are placed through their common EMR) and collects all of the information needed to assess clinical care quality using Healthcare Effectiveness Data and Information Set (HEDIS) measures. Data from this system have been used in numerous prior analyses of healthcare quality.

ELIGIBILITY:
Inclusion Criteria:

• Providers who can place orders in the EMR independently and who have worked at ATRIUS since 2013.

Exclusion Criteria:

• Providers who do not use the common electronic medical record system, cannot place orders in the electronic medical record independently (e.g., registered nurses, licensed practical nurses, registered dieticians), worked after hours Telecom, or were per diem.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Overall procedure and imaging test ordering rate | 1 year
Choosing Wisely-based clinically inappropriate ordering rate | 1 year
HEDIS-based clinically appropriate ordering rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alyna T Chien, MD, MS, Principal Investigator — Assistant Professor of Pediatrics, Department of General Pediatrics, Division of Medicine, Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States